CLINICAL TRIAL: NCT01873625
Title: Resurfacing Articular Cartilage With Mesenchymal Stem Cells Transplantation in Patients With Knee Joint Osteoarthritis Affected by Rheumatoid Arthritis: Randomized Triple Blind Clinical Trial Phase II/III (ACRCT)
Brief Title: Transplantation of Bone Marrow Derived Mesenchymal Stem Cells in Affected Knee Osteoarthritis by Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-RA-001
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
Keywords: mesenchymal stem cells; osteoarthritis; arthritis rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Normal salin injection in patients with rheumatoid arthritis for resurfacing of articular cartilage of knee due to osteoarthritis.
  Interventions: Biological: placebo
- mesencymal stem cell (Active Comparator): Mesenchymal stem cell transplantation in patients with rheumatoid arthritis for resurfacing of articular cartilage of knee due to osteoarthritis.
  Interventions: Biological: mesenchymal cell transplantation

INTERVENTIONS:
Biological: mesenchymal cell transplantation — Mesenchymal stem cell transplantation in patients with rheumatoid arthritis for resurfacing of articular cartilage of knee due to osteoarthritis.
  Arms: mesencymal stem cell
Biological: placebo
  Arms: placebo

SUMMARY:
Osteoarthritis of the knee is one of the most common causes of disability among elderly. Arthritis rheumatoid is an autoimmune disease which causes multi articular arthritis, such as knee osteoarthritis. As the disease progresses the cartilage become frustrated, surrounding bone react to become thicker and inflammation occurs in subchondral bone seen in T2-weighted MRI as increase in signal density. Patients are treated initially by pain management. In patients who don't response to first line treatment invasive treatment like total knee replacement is done. The investigators designed this clinical study with the aim of evaluating therapeutic effects of intra-articular injection of bone marrow mesenchymal stem cells (BM-MSCs) in 60 patients with knee osteoarthritis.

DETAILED DESCRIPTION:
In this study all eligible patients were randomly allocated into two study groups by a permuted block randomization method: group A (control group) received only routine medical therapies and placebo injected into there knees.. Group B received mesenchymal stem cells in addition of routine medical therapy.

Patients were categorized according to the following stimulation protocols:

To assess the outcomes, after mesenchymal stem cells transplantation at months 1,3,6 and 12 we will examine the patients by: WOMAC questioners, DAS28 scoring , radiographies assessments and biochemical analysis with laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Body mass index (BMI) ≤30 kg/m2
3. The presence of osteoarthritis based on MRI and American Rheumatism Association criteria since 6 months before invitation

Exclusion Criteria:

1. Response to routine treatment at last one year.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
pain | 1month
  Evaluation the pain reduction after mesenchymal stem cell transplantation that measured by VAS scaling.
physical activity | 1month
  evaluation the improvement of physical activity after mesenchymal stem cell transplantation that measured by WOMAC scoring.
walking distance | 1month
  Evaluation the walking distance after mesenchymal transplantation.

SECONDARY OUTCOMES:
Imaging | 6months
  Evaluation the resurfacing of articular cartilage after mesenchymal transplantation by MRI and radio logic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of regenerative medicine department, head of Royan cell therapy center; Mohsen Emadedin, MD, Study Director — Royan Institute,Department of regenerative medicine; Farhad gharibdoost, MD, Study Director — President of rheumatologic association center of Iran; Soraya Shadmanfar, MD, Principal Investigator — Royan Institute, Department of regenerative medicine
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Shadmanfar S, Labibzadeh N, Emadedin M, Jaroughi N, Azimian V, Mardpour S, Kakroodi FA, Bolurieh T, Hosseini SE, Chehrazi M, Niknejadi M, Baharvand H, Gharibdoost F, Aghdami N. Intra-articular knee implantation of autologous bone marrow-derived mesenchymal stromal cells in rheumatoid arthritis patients with knee involvement: Results of a randomized, triple-blind, placebo-controlled phase 1/2 clinical trial. Cytotherapy. 2018 Apr;20(4):499-506. doi: 10.1016/j.jcyt.2017.12.009. Epub 2018 Feb 7. PMID 29428486
- See also: Related Info — http://RoyanInstitute.org